CLINICAL TRIAL: NCT06715345
Title: Sponsor-initiated Clinical Study to Evaluate the Efficacy and Safety of Novosis Putty for Bone Fusion in Patients Requiring Posterior Instrumentation and Transforaminal Lumbar Interbody Fusion Due to Degenerative Lumbar Disease
Brief Title: Efficacy and Safety of Novosis Putty for Degenerative Lumbar Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CGBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2201
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Degenerative Lumbar Diseases
Keywords: TLIF; Degenerative lumbar diseases; BMP-2
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: single blind( subject - blind, investigator -open, Outcome assessor- blind)
Who Masked: Participant, Outcomes Assessor
Masking Description: single blind( subject - blind, investigator -open, Outcome assessor- blind)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (No Intervention): Local autologous bone
- Experimental Group 1 (Experimental): Dose 1
  Interventions: Device: Bone graft materials and rhBMP-2
- Experimental Group 2 (Experimental): Dose 2
  Interventions: Device: Bone graft materials and rhBMP-2
- Experimental Group 3 (Experimental): Dose 3
  Interventions: Device: Bone graft materials and rhBMP-2

INTERVENTIONS:
Device: Bone graft materials and rhBMP-2 — NOVOSIS PUTTY is a product composed of recombinant human bone morphogenetic protein-2 and β-tricalcium phosphate/hydrogel complex.
  Arms: Experimental Group 1; Experimental Group 2; Experimental Group 3

SUMMARY:
This clinical study aims to evaluate the efficacy and safety of NOVOSIS PUTTY for bone fusion in patients requiring posterior instrumentation and transforaminal lumbar interbody fusion (TLIF) due to degenerative lumbar disease.

DETAILED DESCRIPTION:
The Subject is a patient requiring posterior instrumentation and transforaminal lumbar interbody fusion (TLIF) due to degenerative lumbar disease.

This clinical study aims to compare and evaluate the efficacy and safety of three dose groups of NOVOSIS PUTTY for bone fusion compared to the autologous bone in patients requiring posterior instrumentation and TLIF in the single level between L2 and S1(L2-S1) due to degenerative lumbar disease.

* Control Group (n=12): Local autologous bone
* Experimental Group 1 (n=12): Dose 1
* Experimental Group 2 (n=12): Dose 2
* Experimental Group 3 (n=12): Dose 3

ELIGIBILITY:
Inclusion Criteria:

* Adult aged ≥ 22 to ≤ 80 years
* Subjects whose skeletal maturation are confirmed by showing the result of Risser stage 5 in Risser classification, the Plain Radiography
* Subjects diagnosed with disc degeneration in the single level (L2-S1) lumbar spine along with spondylolisthesis of Meyerding grade 1 (degree of translocation: 0- <25%) or 2 (degree of translocation: 25- <50%) based on the results of radiological examination (CT, MRI, X-ray).
* Subjects with an ODI (Oswestry Disability Index) score of ≥ 35/100 at screening
* Subjects who were treated with non surgical treatment/therapy for at least 3 months, but were judged to have failed treatment by the investigator
* Subjects who are willing to participate in the study, comply with treatment and procedures, and visit the hospital for all observational evaluations
* Subjects who voluntarily signed the informed consent form after hearing the explanation on objectives and methods of this study

Exclusion Criteria:

* Subjects who have a history of medical device application (spinal instrumentation, for example, anterior disc replacement, interspinous device) to the target site or interbody fusion
* Subjects who are considered that the symptoms occurring in the lumbar region are not occurred by disc degeneration
* Subjects with active malignancy
* Subjects with a documented history of drug abuse (e.g., psychotropic drugs including narcotic analgesics and drugs with high dependence such as alcohol) within the last 6 months
* Subjects with a history of endocrine or metabolic disorders known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehler Danlos disease, or osteogenesis imperfecta)
* Subjects with BMI ≥ 35
* Subjects with spondylolis thesis/retrolisthesis with ≥ Grade 3 in the target level
* Subjects with a local acute infection at the current surgical site or active systemic infection (e.g., viral infections such as AIDS, HIV or hepatitis)
* Subjects with a history of metabolic or endocrine diseases known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers Danlos disease, osteogenesis imperfecta, fibrous dysplasia, etc.)
* Subjects with osteoporosis with a mean lumbar spine T-score of ≤ 2.5 on the DEXA bone density test and with a history of osteoporotic fractures (wrist fractures, femur fractures, lumbar spine fractures, etc.)
* Subjects who need to administer drugs that inhibit bone metabolism within 2 weeks after surgery, or Subjects who need to receive post operative drugs that are expected to interfere with bone fusion, such as steroids
* Subjects who smoke ≥ 20 cigarettes a day
* Subjects with autoimmune disease
* Subjects who were exposed to rhBMP 2 in the past
* Subjects who require to get fusion of two or more vertebral levels
* Subjects who have a pseudoarthrosis after previous fusion
* Subjects who had a history of at least one non fusion spinal surgery on the level to be operated
* Subjects who are considered to have a disease that hinders the accurate evaluation (e.g., neuromuscular disease, serious psychiatric disease) at the discretion of the investigator
* Subjects who are pregnant at screening or who are planning to become pregnant during the study participation period
* Subjects who are currently lactating or who are planning to lactate during the study
* Subjects who participated in studies for other drugs, biologics, or medical devices within 6 months from the date of surgery
* Subjects who are in a difficult situation to comply with study related matters

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall bone fusion rate | 12 months after surgery
  Meet the definition of bone fusion based on CT and the definition of bone fusion based on X-ray simultaneously.
Overall fusion success rate | 12 months after surgery
  Meet all of the following conditions:
  1. Success in ODI
  2. Overall Bone Fusion Success
  3. Neurological Success
  4. No serious adverse event
  5. No re-operation

SECONDARY OUTCOMES:
Overall fusion success rate | 6 and 24 months after surgery
  Meet all of the following conditions:
  1. Success in ODI
  2. Overall Bone Fusion Success
  3. Neurological Success
  4. No serious adverse event
  5. No re-operation
Bone fusion rate | 6, 12, and 24 months after surgery
  Bone fusion rate based on CT, X-ray
Oswestry Disability Index(ODI) | 6 weeks, 3, 6, 12, and 24 months after surgery
  Evaluate Oswestry Disability Index(ODI) score/ lowest 0(best) to highest 50(worst)
SF-12 scores (general condition test) | 6 weeks, 3, 6, 12, and 24 months after surgery
  Evaluate SF-12 scores / lowest 0(worst) to highest 100(best)
Numerical Rating Scale (NRS) | 6 weeks, 3, 6, 12, and 24 months after surgery
  Evaluate Numerical Rating Scale (NRS) scores / lowest 0(best) to highest 30(worst)
Neurological Symptoms | 6 weeks, 3, 6, 12, and 24 months after surgery
  Evaluate Neurological Symptoms test/ check among the 3 questions(Worsened/ Constent/Improved) best is imporved, worst is worsened
Satisfaction rate | 6 weeks, 3, 6, 12, and 24 months after surgery
  Evaluate Satisfaction rate score / lowest 0(worst) to highest 3(best)

CONTACTS AND LOCATIONS:
Overall Officials: Jumi Han, Study Chair — CGBio Inc.
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No